CLINICAL TRIAL: NCT00772473
Title: Correlation of Calcitonin Gene-Related Peptide (CGRP) Levels in Saliva With the Evolution of an Attack of Migraine
Status: Completed | Type: Observational
Sponsor: Clinvest (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Roger K. Cady, M.D., Clinvest, A Division of Banyan Group, Inc
Other Study IDs: Migraine IISP 33467
Record Dates: First submitted 2008-10-13; First posted 2008-10-15 (Estimated); Last update posted 2009-05-25 (Estimated); Status verified 2009-05

CONDITIONS: Headache, Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1 group, usual acute triptan treatment
  Interventions: Other: subjects personal triptan

INTERVENTIONS:
Other: subjects personal triptan — Subjects will treat 1 migraine attack with their usual triptan

SUMMARY:
To assess CGRP levels in saliva through the evolution of migraine.

DETAILED DESCRIPTION:
The release of CGRP is assumed to be initiated early in the migraine process and increases as the headache intensifies. Levels of CGRP will be measured during the premonitory, mild, moderate, and severe phases of a single migraine attack and compared to the baseline value determined when the subject was headache free. Understanding of the clinical evolution of migraine CGRP release may have significant implications in acute treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to read, understand, and sign the informed consent
2. Subject is between the ages of 18 and 65, either male or female
3. Negative pregnancy test for those of childbearing potential.
4. Adequate birth control as approved by the investigator if of childbearing potential
5. Subjects must fulfill criteria for IHS migraine (1.1 or 1.2) with a history of 1-6 migraines per month within the past 3 months and at least 15 headache free days though out the previous three month time period

Exclusion Criteria:

1. Pregnant or breast feeding
2. Presence of any condition or symptoms that would knowingly alter the content of the saliva
3. Presence of any medical disease or condition that would interfere with the conduct of the study
4. Current use of other medications that would be contraindicated in those patients that will take triptan medications for treatment of migraine symptoms, ie. MAO inhibitors, lithium, methyergonovine, methysergide, or ergotamine-containing products
5. Use of migraine preventive medications in the three months prior to screening
6. History of drug or alcohol abuse that would interfere with the study
7. Any pathology of the salivary glands such as sialadenitis (e.g., Sjorgen's syndrome, viral or bacterial sialadenitis, obstructive sialadentitis)
8. History of hypersensitivity or allergy to triptan medications
9. Presence of diabetes, salivary gland tumors, liver disease, alcoholism, and neuropathy
10. More than 15 days per month of headache within the past 3 months
11. Participation in another investigative drug study within the past 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at a mid west headache specialty clinic
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Compare baseline levels of CGRP measured during a migraine free period to those during the 4 phases (prodrome, mild, mod., severe) of migraine. | baseline,prodrome, mild, mod., severe, 4 hrs. post dose

SECONDARY OUTCOMES:
CGRP levels compared to no headache and as function of prodrome symptoms, prediction of mod/sev headache; compare prodrome symptoms to those reported at screening to pre-tx,tx,post tx. | screening, prodrome, pre-treatment, mild, moderate tosevere, post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Roger K Cady, M.D., Principal Investigator — Clinvest
Locations (1):
- Clinvest, Springfield, Missouri, United States

REFERENCES:
- [Derived] Cady RK, Vause CV, Ho TW, Bigal ME, Durham PL. Elevated saliva calcitonin gene-related peptide levels during acute migraine predict therapeutic response to rizatriptan. Headache. 2009 Oct;49(9):1258-66. doi: 10.1111/j.1526-4610.2009.01523.x. PMID 19788468